CLINICAL TRIAL: NCT03948633
Title: Improving the Vaccination Experience at School in Calgary
Brief Title: Feasibility of Implementation of CARD for School-Based Immunizations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Anna Taddio, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 36893
Record Dates: First submitted 2019-04-24; First posted 2019-05-14 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Immunisation Anxiety Related Reaction
Keywords: school vaccinations; pain management; knowledge translation
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: This is a feasibility study including 2 community health centres that have been randomly selected to either the multi-faceted knowledge translation intervention (CARD) or control (standard care) out of 8 community health centres anticipated to participate in a future cluster trial. Within each community health centre, 5 individual schools will be randomly selected to participate.
Who Masked: Participant
Masking Description: Students will not be aware of whether they are in the intervention or control group. Care providers who are trained in the intervention are aware of the group allocation. They will not communicate with care providers not trained in the intervention. Care providers that are trained in the intervention will not deliver care to participants in the control group and care providers that are not trained in the intervention will not deliver care to participants in the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARD (multi-faceted knowledge translation intervention) (Experimental): CARD will be integrated into the school vaccination program. This includes pre-vaccination day preparation (e.g., planning of clinic spaces, student and school staff education about CARD) and vaccination day activities (e.g., clinic set-up, processes for triaging students, implementing pain/fear/fainting mitigation interventions from CARD during vaccination).
  Interventions: Other: Multi-faceted knowledge translation intervention
- Control (No Intervention): There are no specific procedures being undertaken to plan or execute clinics. Usual practices will be instituted (i.e., no education specific to CARD, nor clinic set-up or execution to incorporate interventions for pain, fear or fainting).

INTERVENTIONS:
Other: Multi-faceted knowledge translation intervention — The intervention consists of education of relevant stakeholders of best practices and integration of best practices into the vaccination delivery program
  Other Names: CARD
  Arms: CARD (multi-faceted knowledge translation intervention)

SUMMARY:
A multi-faceted knowledge translation intervention - The CARD (C-Comfort, A-Ask, R-Relax, D-Distract) System - was developed to improve the vaccination experience of students at school. CARD is a framework for delivering vaccinations that is student-centred that promotes coping. This study will examine the feasibility of CARD implementation procedures and measures in the school vaccination program in Calgary, Alberta for use in a larger cluster trial.

DETAILED DESCRIPTION:
Vaccination is estimated to have saved more lives in Canada over the last 50 years than any other single intervention and is considered one of the most important advances in the prevention of disease. One major drawback of vaccination, however, is that the usual route of administration involves a painful needle injection. In students undergoing school-based mass vaccinations, vaccine injections frequently cause sever distress and fainting, with some serious injuries resulting from fainting. Concerns about pain and/or needle fear are also directly responsible for vaccine refusal in this population.

An evidence based clinical practice guideline for mitigating vaccine injection pain, fear and fainting has been developed, however, it is not yet implemented across different school-based vaccination settings and students are not benefiting from the research evidence. In a prior small-scale project, investigators developed and implemented a multi-faceted knowledge translation intervention - The CARD (C-Comfort, A-Ask, R-Relax, D-Distract) System - in some schools in a small public health region in Niagara, Ontario. CARD is a framework for delivering vaccinations that is student-centred and promotes coping. It integrates recommendations from the guideline in two separate components of the vaccination delivery program: 1) pre-vaccination day preparation, and 2) vaccination day activities. Investigators found preliminary evidence of acceptability, appropriateness, satisfaction and clinical effectiveness of CARD when used in grade 7 students in Niagara.

In this study, investigators plan to determine the feasibility of implementing CARD in a diverse and more complex public health region in Calgary, Alberta. Specifically, investigators will determine recruitment rates, adherence to CARD protocol, response rates for questionnaires, acceptability, appropriateness (fit), and satisfaction. The results will inform a future cluster trial.

ELIGIBILITY:
Inclusion Criteria:

* grade 9 student eligible for vaccination at school
* public health staff in community health centre involved in the study
* school staff in a participating school involved in school vaccination program
* parent of a student eligible for vaccination at school

Exclusion Criteria:

* unable to understand and read English

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
percent complete data for student symptom survey | within 5 minutes after vaccination
  proportion of students that fill in questionnaire about their symptoms (fear, dizziness, pain) during vaccination

SECONDARY OUTCOMES:
percent complete data for nurse feedback form | within 5 minutes after vaccination
  proportion of immunizers that fill in questionnaire about interventions used during immunization (e.g., privacy, distraction)
percent of schools recruited | within 1 week of school vaccination clinic
  proportion of schools that participate in the study
percent compliance with CARD (intervention) | within 3 months after vaccination
  proportion of adherence to components of CARD protocol as assessed by CARD implementers using a self-reported checklist. This information will be supplemented with information from focus groups with implementers and study notes, as well as focus groups with other stakeholder groups (students, parents, school staff).
perceived quality of CARD (intervention) program delivery | within 3 months after vaccination
  perceptions of quality of CARD program delivery as reported by CARD implementers (primary targets) using the CARD Global Impression Checklist, individual quality questions (5-point likert scale, higher number represents better outcome). This information will be supplemented with information from focus groups with implementers and study notes, as well as focus groups with other stakeholder groups (secondary targets - school staff, students, parents).
perceived acceptability of CARD (intervention) | within 3 months after vaccination
  perception of acceptability (satisfaction with CARD) by CARD implementers (primary targets) using the CARD Global Impression Checklist, individual acceptability questions (5-point likert scale, higher number represents better outcome). This information will be supplemented with information from focus groups with implementers and study notes, as well as focus groups with other stakeholder groups (secondary targets - school staff, students, parents).

OTHER OUTCOMES:
perceived appropriateness of CARD (intervention) | within 3 months of vaccination
  perception of appropriateness (fit of CARD) by CARD implementers (primary targets) using the CARD Global Impression Checklist, individual appropriateness questions (5-point likert scale, higher number represents better outcome). This information will be supplemented with information from focus groups with implementers and study notes, as well as focus groups with other stakeholder groups (secondary targets - school staff, students, parents).
perceived feasibility of CARD (intervention) | within 3 months of vaccination
  perception of feasibility (extent to which CARD can be carried out) by CARD implementers (primary targets) using the CARD Global Impression Checklist, individual feasibility questions (5-point likert scale, higher number represents better outcome). This information will be supplemented with information from focus groups with implementers and study notes, as well as focus groups with other stakeholder groups (secondary targets - school staff, students, parents).
percent reliability of data collection | within 1 day of activities described (education, immunization day, and nurse feedback)
  proportion of agreement between implementer and observer checklists for aspects of immunization program delivery (i.e., education, immunization day, nurse feedback form)
success of recruitment of secondary targets (school staff, students, parents) for focus groups | within 3 months of vaccination
  proportion of focus groups successfully undertaken with secondary stakeholder targets.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — University of Toronto
Locations (1):
- Alberta Health Services Public Health - Calgary Zone, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

REFERENCES:
- [Derived] Taddio A, Coldham J, Logeman C, McMurtry CM, Little C, Samborn T, Bucci LM, MacDonald NE, Shah V, Dribnenki C, Snider J, Stephens D. Feasibility of implementation of CARD for school-based immunizations in Calgary, Alberta: a cluster trial. BMC Public Health. 2021 Feb 1;21(1):260. doi: 10.1186/s12889-021-10247-4. PMID 33526030